CLINICAL TRIAL: NCT03860272
Title: A Phase 1 Study of AGEN1181, an Fc-Engineered Anti-CTLA-4 Monoclonal Antibody as Monotherapy and in Combination With AGEN2034 (Balstilimab), an Anti-PD-1 Monoclonal Antibody, in Subjects With Advanced Cancer
Brief Title: Fc-Engineered Anti-CTLA-4 Monoclonal Antibody in Advanced Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-800-01
Record Dates: First submitted 2019-02-12; First posted 2019-03-01 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Advanced Cancer; Angiosarcoma; Colorectal Cancer Without Liver Metastases; Endometrial Cancer; Fibrolamellar Carcinoma; Non-small-cell Lung Cancer; Ovarian Cancer; Prostate Cancer
Keywords: Solid Tumors; Advanced Cancer; Open-label; Monotherapy; Combination Therapy; Anti-CTLA-4; Anti-PD-1; Immunotherapy
MeSH Terms: conditions — Hemangiosarcoma; Endometrial Neoplasms; Fibrolamellar hepatocellular carcinoma; Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Prostatic Neoplasms | interventions — Ipilimumab; balstilimab; spartalizumab

STUDY DESIGN:
Intervention Model Description: Dose escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 3-Week Monotherapy (Experimental): 3+3 Dose escalation: botensilimab, every 3 weeks, starting at dose level 0.1 milligrams/kilogram (mg/kg) up to 4 mg/kg, administered intravenously (IV) for up to 2 years.
  Interventions: Drug: Botensilimab
- 6-Week Monotherapy (Experimental): 3+3 Dose escalation: botensilimab, every 6 weeks, starting at dose level 1 mg/kg up to 4 mg/kg, administered IV for up to 2 years.
  Interventions: Drug: Botensilimab
- 6-Week Combination Therapy (Experimental): 3+3 Dose escalation: balstilimab, every 2 weeks, at dose level 3 mg/kg in combination with botensilimab, every 6 weeks, starting at dose level 0.1 mg/kg up to 4 mg/kg, administered IV for up to 2 years. Participants enrolled at sites in the United Kingdom (UK) may have the option for extended treatment. An additional cohort will investigate balstilimab, every 3 weeks, at 450 mg in combination with botensilimab every 6 weeks, at 150 mg, administered IV for up to 2 years.
  Interventions: Drug: Botensilimab; Drug: Balstilimab

INTERVENTIONS:
Drug: Botensilimab — An Fc-engineered anti-CTLA-4 monoclonal antibody
  Other Names: AGEN1181; Anti-CTLA-4
Drug: Balstilimab — A fully human monoclonal anti-PD-1 antibody
  Other Names: AGEN2034; Anti-PD-1
  Arms: 6-Week Combination Therapy

SUMMARY:
This study is an open-label, Phase 1, multicenter study to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamic (PD) profiles of a novel fragment crystallizable (Fc)-engineered immunoglobulin G1 anti-cytotoxic T-lymphocyte antigen 4 (anti-CTLA-4) human monoclonal antibody (botensilimab) monotherapy and in combination with an anti-programmed cell death protein-1 (PD-1) antibody (balstilimab), and to assess the maximum tolerated dose (MTD) in participants with advanced solid tumors. This study will also determine the recommended phase 2 dose (RP2D) of botensilimab monotherapy and in combination with balstilimab.

DETAILED DESCRIPTION:
This Phase 1 study will enroll up to approximately 550 evaluable adult participants with refractory, advanced cancer (solid tumors).

The study will consist of a 3+3 dose escalation. Different dose levels of botensilimab, both monotherapy and in combination with balstilimab, will be evaluated in individual cohorts based upon dose. Each participant will remain in the cohort of the dose level and schedule assigned at study entry. Participants can be replaced for any reason other than a dose-limiting toxicity (DLT). Participants will receive treatment for ≤ 2 years or until progressive disease, unacceptable toxicity, or any criterion for stopping the study drug or withdrawal of trial occurs.

Additionally, the study is intended to further explore the safety, PK, PD, and clinical activity in selected cancer types at dose levels (botensilimab monotherapy and combination therapy with balstilimab) determined as potentially effective. Indications of interest include, but are not limited to, non-small-cell lung cancer, melanoma, endometrial cancer, ovarian cancer, angiosarcoma, colorectal cancer without liver metastases, prostate cancer, and fibrolamellar carcinoma.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the trial, all of the following inclusion criteria must be fulfilled, as no waivers will be permitted:

1. Provision of signed and dated written informed consent prior to any study specific procedures. Participation in pharmacogenomics testing is optional.
2. Histologically or cytologically confirmed diagnosis of metastatic or locally advanced solid tumor for which no standard therapy is available or standard therapy has failed.
3. Measurable disease on imaging based on RECIST 1.1, except for prostate cancer.
4. Life expectancy of ≥ 3 months and Eastern Cooperative Oncology Group performance status of 0 or 1.
5. Adequate organ and bone marrow reserve function, as indicated by the following laboratory values:

   1. Adequate hematological function, defined as absolute neutrophil count ≥ 1.5 × 10^9/liter (L), platelet count ≥ 100 × 10^9/L, and hemoglobin ≥ 8 grams/deciliter without recent transfusion (defined as a transfusion that has occurred within 2 weeks of the hemoglobin measurement).
   2. Adequate liver function, defined as total bilirubin level ≤ 1.5 × institutional upper limit of normal (IULN) (except for participants with Gilbert syndrome who must have a total bilirubin level of ≤ 3.0 × IULN), aspartate aminotransferase ≤ 2.5 × IULN, and alanine aminotransferase ≤ 2.5 × IULN.
   3. Adequate renal function defined as creatinine ≤ 1.5 × IULN or measured or calculated creatinine clearance ≥ 40 milliliters (mL)/minute per institutional standard. Assessment methods should be recorded.
   4. Adequate coagulation, defined as international normalized ratio or prothrombin time ≤ 1.5 × IULN and activated partial thromboplastin time ≤ 1.5 × IULN (unless participant receiving anticoagulant therapy) or stable known coagulopathy with sponsor approval.
6. A sufficient and adequate formalin-fixed paraffin embedded tumor tissue sample (fresh or archival tumor tissue) collected since last treatment and before the first dose from a site not previously irradiated, if clinically feasible.
7. Female participants of childbearing potential must have a negative serum pregnancy test at screening (within 72 hours of first dose of study medication). Non-childbearing potential is defined as 1 of the following:

   1. ≥ 45 years of age and has not had menses for > 1 year and there is no alternative medical cause.
   2. Amenorrheic for > 2 years without a hysterectomy and/or oophorectomy and follicle stimulating hormone value in the postmenopausal range upon pretrial (screening) evaluation.
   3. Status is post-hysterectomy, -oophorectomy, or -tubal ligation.
8. Female participants of childbearing potential must be willing to use highly effective contraceptive measures starting with the Screening visit through 90 days after last dose of study treatment. For the UK only, highly effective contraceptive measures are defined as follows:

   1. Combined (estrogen and progesterone containing) hormonal contraception associated with inhibition of ovulation.

      * Oral
      * Intravaginal
      * Transdermal
   2. Progesterone-only hormonal contraception associated with inhibition of ovulation.

      * Oral
      * Injectable
      * Implantable
   3. Intrauterine device
   4. Intrauterine hormone-releasing system
   5. Bilateral tubal occlusion
   6. Vasectomized partner
   7. Sexual abstinence
9. Male participants with a female partner(s) of childbearing potential must agree to use highly effective contraceptive measures throughout the trial starting with the Screening visit through 90 days after the last dose of study treatment is received. Males with pregnant partners must agree to use a condom (which is not considered "highly effective"); no additional method of contraception is required for the pregnant partner. Note: Abstinence is acceptable if this is the established and preferred contraception method for the participant.

   The following inclusion criteria are in addition to the above criteria. If there are criteria below that differs from above, the below indication-specific criteria take precedence.

   Additional Inclusion Criteria for Angiosarcoma Cohort
10. Histologically or cytologically confirmed diagnosis of metastatic or locally advanced angiosarcoma for which no standard therapy is available or standard therapy has failed.

    Additional Inclusion Criteria for the Hepatocellular Cancer (HCC) Cohort
11. Histologically or cytologically confirmed diagnosis or radiological diagnosis following the guidelines from the American Association for the Study of Liver Diseases of metastatic or locally advanced HCC.
12. Must have progressed while receiving, or following, programmed death-ligand 1 (PD(L)-1)-based therapy.
13. Child-Pugh score of A. Note: Participants on anticoagulant treatment would have an assigned value of 1 point when scoring prothrombin time/international normalized ratio so the overall Child-Pugh score is not adversely affected.
14. Adequate organ and bone marrow reserve function as indicated by the following laboratory values:

    1. Platelet count ≥ 60 × 10^6/cubic millimeter (mm^3) and absolute neutrophil count ≥ 1,000 × 10^6/L are acceptable provided that the investigator assesses these abnormalities as being due to liver disease.
    2. Adequate liver function, defined as aspartate aminotransferase and alanine aminotransferase ≤ 5 × IULN, bilirubin ≤ 2 × IULN.
15. Participants are eligible to enroll if they have non-viral-HCC or if they have hepatitis B (HBV), or hepatitis C virus (HCV) related HCC, defined as follows:

    1. Chronic HBV infection as evidenced by detectable HBV surface antigen or HBV DNA. Participants with chronic HBV infection must be on antiviral therapy and have HBV DNA < 500 international units/mL.
    2. Active or resolved HCV infection as evidenced by detectable HCV RNA or antibody.

    Additional Inclusion Criteria for the Non-Small Cell Lung Cancer (NSCLC) Cohort
16. Histologically or cytologically confirmed diagnosis of metastatic or locally advanced NSCLC for which no standard therapy is available or standard therapy has failed:

    1. Adenocarcinoma or squamous cell carcinoma at the time of enrollment. If other histologies are also present, must be approved by the medical monitor prior to study entry.
    2. For participants without targetable alterations: Prior treatment with anti PD(L)-1-based therapy.
    3. Participants with targetable alterations (for example, estimated glomerular filtration rate, anaplastic lymphoma kinase, Kirsten rat sarcoma virus-single point mutation with a glycine-to-cysteine substitution at codon 12, reactive oxygen species, mesenchymal epithelial transition factor receptor, etc.): must have received or be intolerant of at least one approved targeted therapy.

    Additional Inclusion Criteria for the Prostate Cancer Cohort
17. Diagnosis of metastatic castrate resistant prostate cancer.
18. Must have demonstrated serologic or radiographic progression on or following the most recent therapy in the setting of castrate-level testosterone (< 50 nanograms per mL [ng/mL] and/or maintained on medical/surgical castration throughout) as defined by at least one of the following:

    1. Baseline PSA ≥ 2.0 ng/mL and 2 sequential rises in prostate-specific antigen (PSA) with each rising value being at least 1 week apart.
    2. Progression by RECIST 1.1.
    3. Progression by PCWG3 criteria for bone disease ("2+2" rule) with or without PSA progression.
19. Must maintain castration status defined as serum testosterone < 50 ng/mL. Must be either surgically castrate or on luteinizing hormone-releasing hormone analog for the duration of the study.

    Additional Inclusion Criteria for Breast Cancer
20. Must have received PD-(L)1 therapy if indicated. Note: Premenopausal participants may continue ongoing ovarian suppression on study. Permitted agents are goserelin, triptorelin or analogs.

Exclusion Criteria:

For inclusion in the trial, participant must meet none of the following exclusion criteria, as no waivers will be permitted:

1. Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigation device within 3 weeks of first dose of current study drug.
2. Received prior systemic cytotoxic chemotherapy, biological therapy, radiotherapy, or major surgery within 3 weeks prior to first dose of study drug; for tyrosine kinase inhibitor or similar within 4 × half-life prior to first dose of study drug. A 1-week washout is permitted for palliative radiation to non-central nervous system disease, with Sponsor approval.
3. Participants who have received prior CTLA-4 therapy may be enrolled in selected indications upon agreement with the Sponsor.
4. Persistent toxicity of NCI CTCAE version 5.0 Grade > 1 severity that is related to prior therapy. Note: Sensory neuropathy, hypothyroidism or alopecia of Grade ≤ 2 are acceptable. Other Grade 2 toxicities of prior treatments that are controlled with medication (for example, diabetes or hypertension) may be permitted with sponsor approval.
5. Expected to require any other form of systemic or localized antineoplastic therapy while on trial (including maintenance therapy with another agent, radiation therapy, and/or surgical resection).
6. History of:

   1. Severe (Grade ≥ 3) hypersensitivity reaction to a fully human monoclonal antibodies
   2. Immune-related adverse event requiring treatment with systemic steroids for > 7 days excluding Grade 1 or 2 rash.
   3. Interstitial lung disease or lung disease which may interfere with the assessment of pneumonitis.
   4. Uncontrolled asthma (that is, ≥ 3 features of partly controlled asthma)
   5. Pneumonitis that has required oral or IV corticosteroids.
7. Receiving systemic corticosteroid therapy 1 week prior to the first dose of study drug or receiving any other form of systemic immunosuppressive medication. Note: Corticosteroid use as a premedication for IV contrast allergies/reactions is allowed. Participants who are receiving daily corticosteroid replacement therapy are also an exception to this rule. Daily prednisone at doses of ≤ 7.5 mg or equivalent hydrocortisone dose are examples of permitted replacement therapy. Use of inhaled or topical corticosteroids is permitted.
8. Brain metastases or leptomeningeal metastases with the following exceptions: Note: Brain metastases which have been treated with either surgical resection or stereotactic radio surgery. These participants must be off steroids ≥ 10 days prior to enrollment for the purpose of managing their brain metastases. Repeat brain imaging following surgical resection or stereotactic radiosurgery is not required if their last brain magnetic resonance imaging is within screening window. Note: Untreated isolated brain metastases that are too small for treatment by surgical resection or stereotactic radiosurgery (that is, 1-2 mm) and/or of uncertain etiology are potentially eligible but must be approved by the sponsor.
9. Active or history of autoimmune disease that requires systemic treatment within 2 years of the start of study drug (that is, with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Note: Participants with autoimmune conditions requiring hormone replacement therapy or topical treatments are eligible.
10. Has had an allogeneic tissue/solid organ transplant, except for corneal transplants.
11. Active infection requiring systemic treatment.
12. Known history of human immunodeficiency virus type 1 or 2 antibodies.
13. Known active infection with hepatitis B and/or hepatitis C virus.
14. Clinically significant (that is, active) cardiovascular disease: cerebral vascular accident/stroke or myocardial infarction within 6 months of enrollment, unstable angina, congestive heart failure (New York Heart Association class ≥ II), or serious uncontrolled cardiac arrhythmia requiring medication.
15. History or current evidence of any condition, therapy, any active infections, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating Investigator.
16. Known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the study.
17. Legally incapacitated or has limited legal capacity.
18. Pregnant or breastfeeding.
19. Concurrent malignancy requiring treatment or history of prior malignancy active within 2 years prior to the first dose of study treatment. Exceptions: participants with completely resected prior early-stage basal/squamous cell skin cancer or treated cervical carcinoma in situ.

    The following exclusion criteria are in addition to the above criteria. If there are criteria below that differs from above, the below indication-specific criteria take precedence.

    Additional Exclusion Criteria for the HCC Cohort
20. Received locoregional therapy (for example, transcatheter chemoembolization, radiation, surgery) within 6 weeks or yttrium-90 within 12 weeks.
21. Hepatic encephalopathy within the last 6 months requiring admission or initiation of or intensification of therapy. Participants taking rifaximin/lactulose as encephalopathy prophylaxis are allowed as long as they have not had clinically evident encephalopathy in the past 6 months.
22. Gastro-esophageal varices bleeding in the last 6 months.
23. Ascites requiring paracentesis within the last 3 months. Participants with previous ascites that is managed with stable doses of diuretics and have a Child Pugh score of A are allowed.

    Exclusion Criterion Specific for the UK
24. Hypersensitivity to the active ingredient or any other component of the investigational medicinal products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 499 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence Of Treatment-emergent Adverse Events (TEAEs) | First dose through 90 days following last study dose (up to 2 years)
  TEAEs will include adverse events of special interest, immune-related adverse events, and adverse drug reactions, according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0.
DLT Of Botensilimab | First 28 days of treatment
  DLTs will include any Grade 2 or greater drug related toxicity for all dose groups, according to NCI CTCAE version 5.0 and protocol specifications.
RP2D Of Botensilimab | First dose through 90 days following last study dose
  MTD based on DLT occurrence at DLT period (28 days after first dose) and all TEAEs seen through 90 days following last study dose.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) According To Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1) | First dose through up to 2 years
  Confirmed ORR will be in the analysis population.
ORR According to Prostate Cancer Working Group 3 (PCWG3) | First dose through up to 2 years
  Confirmed ORR will be in the analysis population.
Duration Of Response (DOR) According To RECIST 1.1 | From first dose to first observation of documented disease progression (or death within 12 weeks of last tumor assessment) (up to 2 years)
DOR According to PCWG3 | From first dose to first observation of documented disease progression (or death within 12 weeks of last tumor assessment) (up to 2 years)
Disease Control Rate (DCR) According To RECIST 1.1 | First study dose through 24 weeks
  DCR will include complete response, partial response, and stable disease.
DCR According to PCWG3 | First study dose through 24 weeks
  DCR will include complete response, partial response, and stable disease.
Progression-free Survival (PFS) According To RECIST 1.1 | First study dose to first observation of documented disease progression (or death within 12 weeks of last tumor assessment) (up to 2 years)
  PFS time will be assessed.
PFS According to PCWG3 | First study dose to first observation of documented disease progression (or death within 12 weeks of last tumor assessment) (up to 2 years)
  PFS time will be assessed.
Overall Survival Time | First study dose through up to 3 years
  Duration of survival will be assessed.
Maximum Drug Concentration At Steady-state (Cmax-ss) | First study dose (pre-dose) through 3 months following last study dose (up to 2 years)
  Serum botensilimab concentrations measured throughout the study
Minimum Drug Concentration At Steady-state (Cmin-ss) | First study dose (pre-dose) through 3 months following last study dose (up to 2 years)
  Serum botensilimab concentration measured throughout the study
Area Under The Drug Concentration-time Curve Within Time Span t1 To t2 At Steady-state (AUC(t1-t2)-ss) | First study dose (pre-dose) through 3 months following last study dose (up to 2 years)
  Serum botensilimab concentrations measured throughout the study
Area Under The Drug Concentration-time Curve From Time Zero To Infinity [AUC(0-∞)] | First study dose (pre-dose) through 3 months following last study dose (up to 2 years)
  Serum botensilimab concentrations measured throughout the study
Terminal Elimination Rate Constant (λz) | First study dose (pre-dose) through 3 months following last study dose (up to 2 years)
  Serum botensilimab concentrations measured throughout the study
Terminal Elimination Half-life (t1/2) | First study dose (pre-dose) through 3 months following last study dose (up to 2 years)
  Serum botensilimab concentrations measured throughout the study
Systemic Clearance (CL) | First study dose (pre-dose) through 3 months following last study dose (up to 2 years)
  Serum botensilimab concentrations measured throughout the study
Volume Of Distribution (Vd) | First study dose (pre-dose) through 3 months following last study dose (up to 2 years)
  Serum botensilimab concentrations measured throughout the study
Anti-drug Antibodies (ADAs) | First study dose (pre-dose) through 3 months following last study dose (up to 2 years)
  Serum botensilimab ADAs measured throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Agenus Inc.
Locations (18):
- United States (17):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - The Angeles Clinic & Research Institute, a Cedars-Sinai Affiliate, Los Angeles, California
  - University of Southern California Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA Santa Monica Hematology Oncology, Los Angeles, California
  - Saint John's Cancer Institute, Santa Monica, California
  - University of Colorado, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Providence Portland Cancer Center, Portland, Oregon
  - MD Anderson Cancer Center, Houston, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
- Royal Marsden Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bengala E, Santini D, Picone V. Refractory microsatellite-stable metastatic colorectal cancer: a comparison between botensilimab + balstilimab and current standard of care. Immunooncol Technol. 2025 Nov 28;29:101558. doi: 10.1016/j.iotech.2025.101558. eCollection 2026 Mar. PMID 41502912
- [Derived] Wilky BA, Schwartz GK, Gordon MS, El-Khoueiry AB, Bullock AJ, Henick B, Agulnik M, Singh A, Mahadevan D, Stebbing J, Delepine C, Chand D, Avagyan M, Wu W, Johnson B, Grossman JE, O'Day S, Trent JC, Jones RL, Tsimberidou AM. Botensilimab (Fc-enhanced anti-cytotoxic lymphocyte-association protein-4 antibody) Plus Balstilimab (anti-PD-1 antibody) in Patients With Relapsed/Refractory Metastatic Sarcomas. J Clin Oncol. 2025 Apr 10;43(11):1358-1368. doi: 10.1200/JCO-24-02524. Epub 2025 Jan 27. PMID 39869830
- [Derived] Bullock AJ, Schlechter BL, Fakih MG, Tsimberidou AM, Grossman JE, Gordon MS, Wilky BA, Pimentel A, Mahadevan D, Balmanoukian AS, Sanborn RE, Schwartz GK, Abou-Alfa GK, Segal NH, Bockorny B, Moser JC, Sharma S, Patel JM, Wu W, Chand D, Rosenthal K, Mednick G, Delepine C, Curiel TJ, Stebbing J, Lenz HJ, O'Day SJ, El-Khoueiry AB. Botensilimab plus balstilimab in relapsed/refractory microsatellite stable metastatic colorectal cancer: a phase 1 trial. Nat Med. 2024 Sep;30(9):2558-2567. doi: 10.1038/s41591-024-03083-7. Epub 2024 Jun 13. PMID 38871975